CLINICAL TRIAL: NCT05969483
Title: Validation of a Processed EEG Device (pEEG, Masimo Sedline®) as a Monitoring Tool for the Analgosedation Level in Mechanically Ventilated Critically Ill Children
Brief Title: Validation of a Processed EEG Device for Monitoring Sedation in PICU
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, angela amigoni, Director, Azienda Ospedaliera di Padova
Other Study IDs: AOP2549
Record Dates: First submitted 2023-05-20; First posted 2023-08-01 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Sedation Complication
Keywords: sedation; pediatric intensive care; monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- sedated and ventilated pediatric critical care patients: All sedated and ventilated critically ill patients will be exposed to the Masimo Sedline® sensor. Its pEEG scores, including the PSI, will be registered by the patient primary nurse every 4 hours for the first 5 days of ventilation. At the same time, CBS will be evaluated by a specialized PICU nurse and by a critical-care expert physician, blinded to each other. In case of chemically paralyzed patients, a paralysis holiday will be performed when clinically possible . A CBS will be assessed when the paralytic agents will be considered washed out. The patient's analgosedation strategy and analgosedation protocol will not be standardized but will be decided by the treating physician based on the international recommendations.
  Interventions: Device: pEEG monitoring

INTERVENTIONS:
Device: pEEG monitoring — pEEG monitoring during PICU admission

SUMMARY:
The goal of this prospective observational study is to validate pEEG as a monitoring tool for the analgosedation level in mechanically-ventilated critically ill children, receiving or not-receiving NMBAs. The main question aims to answer is to measure the strength of agreement between pEEG score and Comfort Behavioural Scale (CBS) (goal standard).

Participants will be monitored with pEEG and CBS evaluated during PICU admission. paralysis holiday) by a specialized PICU nurse and by a critical-care expert physician, blinded to each other.

DETAILED DESCRIPTION:
Rationale: The existence of a strong agreement between the two scores will allow us to consider the use of Masimo Sedline® PSI in our routine practice as an additional tool to monitor the analgosedation level of mechanically ventilated critically ill patients, as well as the main tool for chemically paralyzed patients.The final goal of this project is to validate the Masimo Sedline® as a monitoring tool for the analgosedation level in mechanically-ventilated critically ill children, receiving or not-receiving NMBAs.

Specific Aim. To evaluate the strength of agreement between CBS and the Masimo Sedline® PSI in children.

Design: prospective cohort study including all consecutive mechanically ventilated patients receivinganalgosedation admitted to a tertiary-care PICU.

Setting: Tertiary-care Center PICU (Padova University Hospital, Italy). Partecipants: all consecutive patients who will receive mechanical ventilation and consequently analgosedation admitted to our PICU during the study period. Both patients receiving NMBAs and patient not receiving NMBAs will be included (patients with NMBA will be evaluated during a paralysis holiday). Exclusion criteria: patient with skin lesions or other significant traumatic lesions in the area where the Masimo Sedline® sensor need to be applied.

Exposure: All patients will be exposed to the Masimo Sedline® sensor. Its pEEG scores, including the PSI, will be registered by the patient primary nurse every 4 hours for the first 5 days of ventilation. At the same time, CBS will be evaluated by a specialized PICU nurse and by a critical-care expert physician, blinded to each other. In case of CBS discordance between the two operators, a mean will be used for data analysis. In case of chemically paralyzed patients, a paralysis holiday will be performed when clinically possible (ideally twice a day). A CBS will be assessed when the paralytic agents will be considered washed out, i.e. when the patient starts triggering at the ventilator and the EMG index starts showing muscular activity. The patient's analgosedation strategy and analgosedation protocol will not be standardized but will be decided by the treating physician based on the international recommendations.

Main outcome and measures: To evaluate the strength of agreement between the Masimo Sedline® PSI (exposure) and the CBS in mechanically in mechanically ventilated children, adequately or inadequately sedated, and in patients receiving NMBAs (during paralysis holiday).

Analytical plan: Descriptive statistics will be used to describe patients' demographic and clinical characteristics, as well as patient-related clinical outcomes. PSI and CBS will be tested for agreement using K statistics separately in patients with adequate sedation (CBS 11-22), inadequate sedation (CBS <11 or >22), and in patients receiving NMBAs. Multiple sensitivity analyses will be also performed in different subcohort of patients, including neonates, patients with seizures, as well as for different drugs. As an additional analysis, the use of a composite score including the EMG index (i.e. muscular activity) and the EEG suppression ratio (measure of EGG suppression events as index of oversedation) will be included.

ELIGIBILITY:
Inclusion Criteria:

- sedated and ventilated patients admitted in PICU

Exclusion Criteria:

* skin lesions
* significant traumatic lesions in the area where the Masimo Sedline® sensor need to be applied.

Ages: 1 Day to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients admitted in PICU who undergone sedation and mechanical (invasive and non invasive) ventilation
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
agreement between PSI (exposure) and CBS scale the CBS | T1 (after 4 hours of ventilation)
  grade of agreement (Kappa of Cohen)
agreement between PSI (exposure) and CBS scale | T1 (after 8 hours of ventilation)
  grade of agreement (Kappa of Cohen)

CONTACTS AND LOCATIONS:
Overall Officials: angela amigoni, MD, Principal Investigator — University Hospital of Padova
Locations (1):
- University Hospital of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Harris J, Ramelet AS, van Dijk M, Pokorna P, Wielenga J, Tume L, Tibboel D, Ista E. Clinical recommendations for pain, sedation, withdrawal and delirium assessment in critically ill infants and children: an ESPNIC position statement for healthcare professionals. Intensive Care Med. 2016 Jun;42(6):972-86. doi: 10.1007/s00134-016-4344-1. Epub 2016 Apr 15. PMID 27084344
- [Result] Amigoni A, Mozzo E, Brugnaro L, Gentilomo C, Stritoni V, Michelin E, Pettenazzo A. Assessing sedation in a pediatric intensive care unit using Comfort Behavioural Scale and Bispectral Index: these tools are different. Minerva Anestesiol. 2012 Mar;78(3):322-9. PMID 22127309
- [Result] Twite MD, Zuk J, Gralla J, Friesen RH. Correlation of the Bispectral Index Monitor with the COMFORT scale in the pediatric intensive care unit. Pediatr Crit Care Med. 2005 Nov;6(6):648-53; quiz 654. PMID 16276329
- [Result] Tobias JD, Grindstaff R. Bispectral index monitoring during the administration of neuromuscular blocking agents in the pediatric intensive care unit patient. J Intensive Care Med. 2005 Jul-Aug;20(4):233-7. doi: 10.1177/0885066605276806. PMID 16061906
- [Result] Christenson C, Martinez-Vazquez P, Breidenstein M, Farhang B, Mathews J, Melia U, Jensen EW, Mathews D. Comparison of the Conox (qCON) and Sedline (PSI) depth of anaesthesia indices to predict the hypnotic effect during desflurane general anaesthesia with ketamine. J Clin Monit Comput. 2021 Dec;35(6):1421-1428. doi: 10.1007/s10877-020-00619-3. Epub 2020 Nov 19. PMID 33211251
- [Result] Ista E, van Dijk M, Tibboel D, de Hoog M. Assessment of sedation levels in pediatric intensive care patients can be improved by using the COMFORT "behavior" scale. Pediatr Crit Care Med. 2005 Jan;6(1):58-63. doi: 10.1097/01.PCC.0000149318.40279.1A. PMID 15636661
- [Result] Smith HAB, Besunder JB, Betters KA, Johnson PN, Srinivasan V, Stormorken A, Farrington E, Golianu B, Godshall AJ, Acinelli L, Almgren C, Bailey CH, Boyd JM, Cisco MJ, Damian M, deAlmeida ML, Fehr J, Fenton KE, Gilliland F, Grant MJC, Howell J, Ruggles CA, Simone S, Su F, Sullivan JE, Tegtmeyer K, Traube C, Williams S, Berkenbosch JW. 2022 Society of Critical Care Medicine Clinical Practice Guidelines on Prevention and Management of Pain, Agitation, Neuromuscular Blockade, and Delirium in Critically Ill Pediatric Patients With Consideration of the ICU Environment and Early Mobility. Pediatr Crit Care Med. 2022 Feb 1;23(2):e74-e110. doi: 10.1097/PCC.0000000000002873. PMID 35119438